CLINICAL TRIAL: NCT00934661
Title: Low Dose Extended-release Epidural Morphine in Conjunction With Lumbar Plexus Block Versus Lumbar Plexus Block Alone for Total Hip Resurfacing Arthroplasty: A Randomized Controlled Trial.
Brief Title: Low Dose Extended-release Epidural and Lumbar Plexus Block Compared to Lumbar Plexus Block for Total Hip Resurfacing
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Drug was discontinued by manufacturer
Sponsor: Wake Forest University (Other)
Collaborators: EKR Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00006969
Record Dates: First submitted 2009-07-02; First posted 2009-07-08 (Estimated); Results first posted 2018-01-16 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Hip Arthroplasty
Keywords: hip resurfacing; hip arthroplasty
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Extended Release Epidural Morphine (Experimental): Four mg (0.4 ml) of EREM will be delivered to the epidural space and flushed with 1 ml of saline
  Interventions: Drug: Extended Release Epidural Morphine (EREM)
- Placebo Group (Placebo Comparator): The epidural injection will be a placebo consisting of 0.4 ml of saline followed by 1 ml saline flush
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Extended Release Epidural Morphine (EREM) — A single Four mg (0.4 ml)dose of EREM will be administered into the epidural space and flushed with 1 ml of saline
  Other Names: Depodur
  Arms: Extended Release Epidural Morphine
Drug: Placebo — A single epidural injection will be a placebo consisting of 0.4 ml of saline followed by 1 ml saline flush
  Other Names: preservative free normal saline; sodium chloride
  Arms: Placebo Group

SUMMARY:
At Wake Forest University, the investigators have been using Extended Release Epidural Morphine (EREM), since late 2004, as part of multimodal analgesia in patients having gynecologic surgeries and hip arthroplasties.

Hypothesis:

In patients undergoing a Birmingham total hip arthroplasty (BHA), low dose EREM in conjunction with lumbar plexus block (LPB) will be better than lumbar plexus block alone in increasing proportion of patients who meet discharge criteria within 24 hours.

DETAILED DESCRIPTION:
Extended release epidural morphine (EREM, DepoDur®: Endo Pharmaceuticals, Chadds Ford PA) has been studied and increasingly utilized as a method to allow for the improved post-operative analgesia of epidural analgesia without infusions.

At Wake Forest University, the investigators have been using EREM, since late 2004, as part of multimodal analgesia in patients having gynecologic surgeries and hip arthroplasties. The investigators initially decreased our dosages from those recommended (15 mg for lower extremity surgery and 10-15 mg for abdominal surgery), because side effects (nausea, vomiting and hypotension) were felt to be limiting to recovery. The investigators now use 4-7.5 mg in most patients, with 7.5 mg being the exception and have achieved better results. For hip arthroplasties, the investigators currently use 4-5 mg and have performed two retrospective chart reviews on this use; both suggesting that this approach is efficacious. However, these doses have not been studied in a prospective, randomized, double blind trial. The investigators would like to evaluate the efficacy of this dose of EREM used as part of a multimodal regimen. The investigators will compare EREM 4 mg with lumbar plexus block versus lumbar plexus block alone, (providing the rest of our multimodal approach for both patients).

ELIGIBILITY:
Inclusion Criteria:

* A primary unilateral Birmingham hip arthroplasty
* Men and women 18-65 years

Exclusion Criteria:

* Refusal of regional anesthesia
* Laboratory evidence of coagulopathy (platelet count less than 100,000 cells/microliter of blood, prothrombin time greater than 12.1 seconds, partial thromboplastin time greater than 30 seconds, or international normalized ratio of greater than 1.5)
* Allergy to morphine
* Obstructive sleep apnea
* Body mass index (BMI) greater than 40 kg/m2
* Pregnant or lactating
* Severe renal or hepatic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela C Nagle, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Extended Release Epidural Morphine | Placebo Group
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Failure of Combined/Spinal Epidural | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended Release Epidural Morphine | Placebo Group | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 11 | 13 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay After Surgery
Time Frame: From surgery day to hospital discharge, up to 4 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Extended Release Epidural Morphine | Placebo Group
Number analyzed (Participants) | 19 | 20
Days | 2.26 (1.29) | 2.51 (2.02)

2. Secondary Outcome: Total Opioid Consumption
Description: Postoperatively, the patients were observed in the post anesthesia care unit (PACU) until regression of sensory levels is demonstrated. They were provided an intravenous (IV) Patient Controlled Analgesia (PCA) and instructions in its use. Morphine 1mg/ml at standard PCA settings (1.5 ml dose, 10 minute lockout interval, 6 ml hourly limit, no basal infusion) were used for postoperative analgesia until discharge plans were made. (Morphine doses were increased in 0.5ml dose increments if the patients were not achieving adequate analgesia.)
Time Frame: 96 hours
Population: Data not collected on Extended Release Epidural Morphine group
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Extended Release Epidural Morphine | Placebo Group
Number analyzed (Participants) | 0 | 20
mg |  | 10.5 (1.8)

3. Secondary Outcome: Patient Satisfaction Score
Description: Verbal satisfaction scores (0-10), higher scores represent better outcomes. Scores will be obtained from patients for 96 hours after surgery.
Time Frame: 96 hours
Population: 17 participants in the Extended Release Epidural Morphine group and 18 participants in the placebo group provided Verbal satisfaction scores
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extended Release Epidural Morphine | Placebo Group
Number analyzed (Participants) | 17 | 18
units on a scale
  Total Mean and Standard Deviation | 9.03 (1.46) | 8.58 (1.49)
  Post Day 1 Surgery: number analyzed (Participants) | 16 | 15
  Post Day 1 Surgery | 9.12 (1.73) | 8.53 (1.28)
  Post Day 2 Surgery: number analyzed (Participants) | 16 | 14
  Post Day 2 Surgery | 8.76 (1.68) | 8.94 (1.29)
  Post Day 3 Surgery: number analyzed (Participants) | 16 | 16
  Post Day 3 Surgery | 9.06 (1.20) | 8.33 (1.57)
  Post Day 4 Surgery: number analyzed (Participants) | 16 | 13
  Post Day 4 Surgery | 9.18 (1.24) | 8.56 (1.82)

4. Secondary Outcome: Distance Walked at Walking Test
Description: Distance walked at walking test. Longer distance walked represent better outcomes
Time Frame: 96 hours
Population: Different amount of observations were different at each visit. Data for Post Surgery Day 4 for the "Extended Release Epidural Morphine" was not collected.
Measure: Mean (Standard Deviation); unit: Steps
Arm/Group | Extended Release Epidural Morphine | Placebo Group
Number analyzed (Participants) | 18 | 20
Steps
  Post Surgery Day 1: number analyzed (Participants) | 16 | 19
  Post Surgery Day 1 | 168.1 (164.2) | 109.8 (117.9)
  Post Surgery Day 2: number analyzed (Participants) | 9 | 12
  Post Surgery Day 2 | 206.7 (97.1) | 143.5 (97.4)
  Post Surgery Day 3: number analyzed (Participants) | 2 | 6
  Post Surgery Day 3 | 200.0 (70.7) | 175.0 (132.8)
  Post Surgery Day 4: number analyzed (Participants) | 0 | 2
  Post Surgery Day 4 |  | 100.0 (141.2)

5. Secondary Outcome: Verbal Pain Scores Post-gait
Description: Verbal pain scores (0-10), lower scores represent better outcomes. Score will be obtained from patients for 1 day after surgery, post gait active and at rest.
Time Frame: 1 day post surgery
Population: 16 participants were analyzed in both the Extended Release Epidural Morphine and the Placebo Group for active pain scores. 17 participants overall were analyzed for the Extended Release Epidural Morphine and 18 participants overall were analyzed for the Placebo Group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extended Release Epidural Morphine | Placebo Group
Number analyzed (Participants) | 17 | 18
units on a scale
  Pain Score Active: number analyzed (Participants) | 16 | 16
  Pain Score Active | 3.44 (2.94) | 7.16 (2.13)
  Pain Score at Rest | 2.35 (2.5) | 3.58 (2.41)

6. Secondary Outcome: Verbal Pain Scores Post-gait
Description: as for outcome 5
Time Frame: 2 Days Post Surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extended Release Epidural Morphine | Placebo Group
Number analyzed (Participants) | 17 | 17
units on a scale
  Pain Score Active | 5.29 (2.23) | 5.24 (2.28)
  Pain Score at Rest | 2.35 (1.41) | 2.41 (1.58)

7. Secondary Outcome: Verbal Pain Scores Post-gait
Description: as for outcome 5
Time Frame: 3 Days Post Surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extended Release Epidural Morphine | Placebo Group
Number analyzed (Participants) | 17 | 18
units on a scale
  Pain Score Active | 4.18 (2.48) | 5.06 (2.29)
  Pain Score at Rest | 2.59 (2.29) | 2.78 (2.05)

8. Secondary Outcome: Verbal Pain Scores Post-gait
Description: as for outcome 5
Time Frame: 4 Days Post Surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extended Release Epidural Morphine | Placebo Group
Number analyzed (Participants) | 17 | 16
units on a scale
  Pain Score Active | 3.59 (2.15) | 5.00 (2.56)
  Pain Score at Rest | 1.88 (2.26) | 2.94 (2.32)

ADVERSE EVENTS:
Arm/Group | Extended Release Epidural Morphine | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Release Epidural Morphine (N=20) | Placebo Group (N=20)
Hypotension (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Subject experienced hypotension during the operative period, continued to experience hypotension during the immediate recovery period and continued on the neosynephrine infusion as well as receiving blood products and colloids for fluid resuscitation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes